CLINICAL TRIAL: NCT03493958
Title: Pilot RCT of Web-based Behavioral Sleep Intervention for Individuals With Alcohol Use Disorder
Brief Title: RCT of Web-Based Behavioral Sleep Intervention for Individuals With Alcohol Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: University of Pennsylvania (Other); University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 180079; 18-CC-0079
Record Dates: First submitted 2018-04-10; First posted 2018-04-11 (Actual); Results first posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2022-09-28

CONDITIONS: Alcohol Use Disorder; Alcohol Dependence; Insomnia
Keywords: Alcohol Dependence; Alcohol Use Disorder; Insomnia; CBTI; Internet CBTI
MeSH Terms: conditions — Alcoholism; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility and acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I (Experimental): Individuals with alcohol use disorder (AUD) in recovery with insomnia completed six online classes that include interactive educational content and case studies about insomnia and its precipitating factors. These sessions are designed to parallel traditional (in-person) cognitive behavioral therapy for insomnia (CBT-I) sessions and are tracked and customized. New sessions are available seven days after completion of the previous session. The program includes a variety of interactive features, including goal setting, feedback based on user-identified symptoms, animations, quizzes, vignettes, and video-based expert explanations. Participants have maximum of 9-11 weeks to complete the six sessions.
  Interventions: Behavioral: Sleep Healthy Using the Internet (SHUTi)

INTERVENTIONS:
Behavioral: Sleep Healthy Using the Internet (SHUTi) — The SHUTi program is an automated, interactive, internet-based intervention based on well-established face-to-face cognitive behavioral therapy for insomnia (CBT-I) components including sleep restriction, stimulus control, sleep hygiene, cognition

SUMMARY:
Background:

Many people with alcohol use disorders have a sleep problem called insomnia. One treatment is Cognitive Behavioral Therapy for Insomnia (CBT-I). Researchers want to study adults experiences with a web-based CBT-I program called SHUTi.

Objective:

To test if a web-based insomnia therapy program works well and helps people with alcohol use disorders.

Eligibility:

Adults ages 18-65 who joined another protocol and have been an inpatient on that protocol at least 14 days.

Design:

Participants will be screened with questions about insomnia. They will wear a device on their wrist and finger for one night while sleeping. This checks for sleep apnea.

Participants will complete 1 of 2 programs:

1. SHUTi: Participants will start using the program in the hospital and finish it about 6 weeks later. They will get a computer tablet to access SHUTi at least 3 times a week. They will get surveys, stories, videos, and interactive data about sleep. They will complete at least 5 daily sleep diaries every week. SHUTi will be customized based on the diaries.
2. Education-only program: This is like SHUTi but it is not interactive and is not customized. Participants will access it at least once a week. They will finish at their own pace within 6 weeks. These participants may access SHUTi later.

All participants will wear a device on their wrist for 4 straight days at several different time points. It records activity and sleep data. They will do this 3 times.

Participants will answer questions about the program before starting it and after finishing. Interviews will be audio recorded.

Participants will do follow-up surveys 6-7 months after they are discharged from the hospital.

DETAILED DESCRIPTION:
Alcohol use disorder (AUD) is characterized by problematic drinking that becomes severe. The prevalence of insomnia in individuals with alcohol dependence is estimated to be between 36-91% and after two weeks of alcohol detoxification, as many as 65% of these individuals still experience "sleep problems." Cognitive behavioral therapy for insomnia (CBT-I) is an efficacious non-pharmacological treatment for insomnia and is recommended as a first-line treatment for adults with chronic insomnia disorder. CBT-I has been associated with more rapid and "durable" improvement in sleep outcomes, even when compared with other nonpharmacological treatments. Internet-based CBT-I (ICBT-I or eCBT-I for "electronic") could play a key role in the dissemination of this behavioral sleep intervention, given the paucity of trained clinicians able to provide CBT-I in person and other logistical/cost concerns. SHUTi (Sleep Healthy Using The Internet) is the most tested and empirically-sound internet intervention for insomnia. The SHUTi program tailors specific recommendations based on participant responses to sleep diaries and other input within the program. Despite the promise of internet-based CBT-I interventions, very little is known about their effectiveness among individuals with AUD: to date, no RCTs exist examining the feasibility/effectiveness of an internet-based CBT-I program among individuals recovering from AUD. This is a two-phase randomized controlled trial assessing feasibility/acceptability and effectiveness of the SHUTi program for research participants at the NIH Clinical Center. Phase I will be focused on assessing feasibility and effectiveness of program delivery and data collection (n=10). Phase II will be a pilot RCT powered to examine intervention effectiveness (n=20 per group). All participants enrolled in this study will first be admitted under the screening and assessment protocol on the 1SE clinic (14-AA-0181), which includes adults over 18 years of age seeking treatment for alcohol rehabilitation. Participants for this study must also meet criteria for "mild to severe" insomnia. Individuals randomized to the intervention group will receive six sessions of the SHUTi intervention (one completed while inpatient, the rest while outpatient) and individuals randomized to the control group will receive an educational web-based program. The goals of the study are as follows: 1) assess the feasibility and acceptability of Internet-based CBT-I among individuals with AUD in recovery with insomnia (Phase I ), 2) compare the efficacy of CBT-I versus control group with respect to primary and secondary outcome variables (Phase II), and 3) explore specific domains associated with improved outcomes: e.g. demographic, psychiatric, and/or drinking-related factors (Phase II). Primary outcome measures include changes in insomnia severity over time and changes in actigraphy-recorded sleep efficiency over time.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants will be eligible for this study if they:

* Are 18-65 years old
* A score of 10 or higher on the Insomnia Severity Index*
* Are admitted as a treatment-seeking inpatient on 1SE under protocol 14-AA-0181 (signing both the clinical and research consent)
* Have been inpatient for at least 14 days prior to consent/screening
* Can speak, understand, and write in English
* Are able to comply with study requirements (including ability to access the Internet at least 2x per week)

EXCLUSION CRITERIA:

Participants will be ineligible for this study if they:

* Are pregnant
* Are a prisoner
* Report a physician diagnosis of moderate to severe obstructive sleep apnea (OSA) OR test positive for moderate to severe OSA as documented with an Apnea Hypopnea Index of 15 events/hour based on WatchPAT testing results
* Have irregular sleep schedules that prevent the ability to follow treatment recommendations (i.e. usual bedtimes outside of 8:00 pm to 2:00 am or arising times outside of 4:00 am to 10:00 am)
* Meet SCID-5/DSM-5 criteria for opioid use disorder in the past year
* Meet SCID-5/DSM-5 criteria for severe cocaine use disorder and/or severe cannabis use disorder in the past year
* Meet diagnostic criteria for an unstable or serious psychiatric condition (schizophrenia, bipolar, major depressive disorder not currently in remission) - based on diagnosis from the SCID for DSM-5
* Are participating in any experimental pharmacological intervention study
* Presence of unstable or serious medical/neurologic illness at PI and MAI discretion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gwenyth R Wallen, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-CC-0079.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nine consented participants did not start the study. 8 of the 9 consented participants were screen failure and one withdrew prior to start of study procedures
Groups:
- Feasibility and Effectiveness of Sleep Healthy Using the Internet (SHUTi) for CBT-I: Individuals with alcohol use disorder (AUD) in recovery with insomnia completed six online classes that include interactive educational content and case studies about insomnia and its precipitating factors. These sessions are designed to parallel traditional (in-person) cognitive behavioral therapy for insomnia (CBT-I) sessions and are tracked and customized. New sessions are available seven days after completion of the previous session. The program includes a variety of interactive features, including goal setting, feedback based on user-identified symptoms, animations, quizzes, vignettes, and video-based expert explanations. Participants have maximum of 9-11 weeks to complete the six sessions.
Period: Overall Study
Arm/Group | Feasibility and Effectiveness of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Started | 25
Completed | 10
Not Completed | 15
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 7
Not completed — Did not complete all required study procedures | 2

BASELINE CHARACTERISTICS:
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 12
  More than one race | 2
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Internet Evaluation and Utility Questionnaire: Average Number of Log in to SHUTi Per Week During the Last 9 Weeks
Description: Average number of times participants logged into SHUTi 9-11 weeks after SHUTi initiation was measured using a survey item, "On average, how many times did you log in to SHUTi per week during the last 8-9 weeks?"
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Evaluation and Utility Questionnaire
Measure: Mean (Standard Deviation); unit: logins per week
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
logins per week | 6 (1.07)

2. Primary Outcome: Internet Evaluation and Utility Questionnaire: Average Time Spent on SHUTi After Logging in
Description: Average amount of time (in minutes) participants spent on SHUTi in the last 9-11 weeks was measured using a survey item, "When you logged in, on average, how much time did you spend on SHUTi?"
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Evaluation and Utility Questionnaire
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Minutes | 14.9 (9.83)

3. Primary Outcome: Internet Evaluation and Utility Questionnaire: Participants With Technical Difficulties Using SHUTi or Tablet
Description: Participants expressed technical difficulties with SHUTi or study provided tablet using a survey item, "Did you have technical difficulties with SHUTi or your tablet?" with a "yes or no" response
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Evaluation and Utility Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = No | 8
  1 = Yes | 3

4. Primary Outcome: Internet Evaluation and Utility Questionnaire: Participants Response to "How Comfortable Are You Using the Handheld Tablet?"
Description: Participants expressed comfort using the tablet with a survey item on a 5-point scale, "How comfortable are you using the handheld tablet?" with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Evaluation and Utility Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not at all | 0
  1 = Slightly | 0
  2 = Somewhat | 0
  3 = Mostly | 0
  4 = Very | 11

5. Primary Outcome: Internet Evaluation and Utility Questionnaire: Participants Response to "How Easy Was SHUTi to Use?"
Description: Participants ease of using SHUTi was measured with a survey item on a 5-point scale, "How easy was SHUTi to use?" with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Evaluation and Utility Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not at all | 0
  1 = Slightly | 0
  2 = Somewhat | 0
  3 = Mostly | 1
  4 = Very | 10

6. Primary Outcome: Internet Evaluation and Utility Questionnaire: Participants Response to "How Convenient Was SHUTi to Use?"
Description: Participants expressed convenience of using SHUTi with a survey item on a 5-point scale, "How convenient was SHUTi to use?" with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Evaluation and Utility Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not at all | 0
  1 = Slightly | 0
  2 = Somewhat | 2
  3 = Mostly | 1
  4 = Very | 8

7. Primary Outcome: Internet Evaluation and Utility Questionnaire: Participants Response to "Extent of SHUTi Keeping Their Interest and Attention"
Description: Participants expressed extent of SHUTi keeping their interest and attention with a survey item on a 5-point scale, "How much did SHUTi keep your interest and attention?" with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Evaluation and Utility Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not at all | 0
  1 = Slightly | 0
  2 = Somewhat | 4
  3 = Mostly | 6
  4 = Very | 1

8. Primary Outcome: Internet Evaluation and Utility Questionnaire: Participants Response to "SHUTi Likeability"
Description: Participants expressed SHUTi likeability with a survey item on a 5-point scale, "How much did you like SHUTi?" with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Evaluation and Utility Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not at all | 0
  1 = Slightly | 1
  2 = Somewhat | 4
  3 = Mostly | 2
  4 = Very | 4

9. Primary Outcome: Internet Evaluation and Utility Questionnaire: Participants Response to "SHUTi Appearance Likeability"
Description: Participants expressed SHUTi appearance likability with a survey item on a 5-point scale, "How much did you like the way SHUTi looked?" with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Evaluation and Utility Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not at all | 0
  1 = Slightly | 0
  2 = Somewhat | 0
  3 = Mostly | 3
  4 = Very | 8

10. Primary Outcome: Internet Evaluation and Utility Questionnaire: Participants Response to "SHUTi Privacy Concerns"
Description: Participants expressed SHUTi privacy concerns with a survey item on a 5-point scale, "How worried were you about your privacy when using SHUTi?" with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Evaluation and Utility Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not at all | 9
  1 = Slightly | 0
  2 = Somewhat | 0
  3 = Mostly | 1
  4 = Very | 1

11. Primary Outcome: Internet Evaluation and Utility Questionnaire: Participants Response to "SHUTi Satisfaction"
Description: Participants expressed satisfaction with SHUTi with a survey item on a 5-point scale, "How satisfied were you with SHUTi?" with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Evaluation and Utility Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not at all | 0
  1 = Slightly | 0
  2 = Somewhat | 2
  3 = Mostly | 1
  4 = Very | 8

12. Primary Outcome: Internet Evaluation and Utility Questionnaire: Participants Response to "Usefulness of SHUTi Information"
Description: Participants expressed usefulness of SHUTi information with a survey item on a 5-point scale, "How useful did you find the information in SHUTi?" with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Evaluation and Utility Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not at all | 0
  1 = Slightly | 0
  2 = Somewhat | 1
  3 = Mostly | 1
  4 = Very | 9

13. Primary Outcome: Internet Evaluation and Utility Questionnaire: Participants Response to "Understanding SHUTi Information"
Description: Participants expressed how easy the SHUTi information was to understand with a survey item on a 5-point scale, "How easy is the information to understand?" with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Evaluation and Utility Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not at all | 0
  1 = Slightly | 0
  2 = Somewhat | 0
  3 = Mostly | 2
  4 = Very | 9

14. Primary Outcome: Internet Evaluation and Utility Questionnaire: Participants Response to "Trust in SHUTi Information Provided"
Description: Participants expressed how well they trusted the SHUTi information provided with a survey item on a 5-point scale, "How much did you feel you could trust the information?" with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Evaluation and Utility Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not at all | 0
  1 = Slightly | 0
  2 = Somewhat | 0
  3 = Mostly | 3
  4 = Very | 8

15. Primary Outcome: Internet Evaluation and Utility Questionnaire: Participants Likelihood of Continued SHUTi Use When Sleep Problems Continue or Return
Description: Participants expressed their likelihood of continued SHUTi when sleep problems continue or return with a survey item on a 5-point scale, "If sleep difficulties were to continue or return, how likely would you be to continue to use SHUTi?" with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Evaluation and Utility Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not at all | 0
  1 = Slightly | 1
  2 = Somewhat | 1
  3 = Mostly | 4
  4 = Very | 5

16. Primary Outcome: Internet Evaluation and Utility Questionnaire: Participants Likelihood of Continued SHUTi Use Due to Technical Difficulties
Description: Participants expressed their likelihood of continued SHUTi if technical difficulties continued with a survey item on a 5-point scale, "If technical difficulties were to continue or return, how likely would you be to continue to use SHUTi?" with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Evaluation and Utility Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not at all | 0
  1 = Slightly | 1
  2 = Somewhat | 3
  3 = Mostly | 3
  4 = Very | 4

17. Primary Outcome: Internet Evaluation and Utility Questionnaire: Participants Response to "Internet as a Delivery Method for Insomnia Intervention"
Description: Participants expressed their feedback regarding delivering insomnia intervention using the internet with a survey item on a 5-point scale, "How good of a method was the Internet for providing this information?" with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Evaluation and Utility Questionnaire. One of 11 participants who completed this questionnaire did not respond to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 10
Participants
  0 = Not at all | 0
  1 = Slightly | 0
  2 = Somewhat | 2
  3 = Mostly | 1
  4 = Very | 7

18. Primary Outcome: Internet Impact and Effectiveness Questionnaire: Participants Response to "SHUTi Helpfulness"
Description: Participants expressed how helpful SHUTi was with a survey item on a 5-point scale, "SHUTi was helpful" with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Impact and Effectiveness Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not at all | 0
  1 = Slightly | 0
  2 = Somewhat | 1
  3 = Mostly | 3
  4 = Very | 7

19. Primary Outcome: Internet Impact and Effectiveness Questionnaire: Participants Response to "Increase in Insomnia Knowledge"
Description: Participants expressed how their insomnia knowledge increased with a survey item on a 5-point scale, "My knowledge about insomnia increased" with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Impact and Effectiveness Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not at all | 0
  1 = Slightly | 0
  2 = Somewhat | 0
  3 = Mostly | 3
  4 = Very | 8

20. Primary Outcome: Internet Impact and Effectiveness Questionnaire: Participants Response to "Quality of Life Improvement"
Description: Participants expressed any quality of life improvement as a result of SHUTi with a survey item on a 5-point scale, "SHUTi improved my overall quality of life" with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Impact and Effectiveness Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not at all | 1
  1 = Slightly | 0
  2 = Somewhat | 4
  3 = Mostly | 2
  4 = Very | 4

21. Primary Outcome: Internet Impact and Effectiveness Questionnaire: Participants Response to "Mood Improvement"
Description: Participants expressed any mood improvement as a result of SHUTi with a survey item on a 5-point scale, "SHUTi helped improve my overall mood" with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Impact and Effectiveness Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not at all | 0
  1 = Slightly | 0
  2 = Somewhat | 3
  3 = Mostly | 4
  4 = Very | 4

22. Primary Outcome: Internet Impact and Effectiveness Questionnaire: Participants Response to "Physical Activity Improvement"
Description: Participants expressed any physical activity improvement (e.g. exercise or sports activities) as a result of SHUTi with a survey item on a 5-point scale, "SHUTi helped improve my level of physical activities, such as exercise regimen or sports activities" with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Impact and Effectiveness Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not at all | 3
  1 = Slightly | 0
  2 = Somewhat | 5
  3 = Mostly | 0
  4 = Very | 3

23. Primary Outcome: Internet Impact and Effectiveness Questionnaire: Participants Response to "Ability to Manage Insomnia"
Description: Participants expressed any increased effectiveness in the ability to manage insomnia as a result of SHUTi with a survey item on a 5-point scale, "SHUTi helped me feel more sure of my ability to manage my insomnia" with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Impact and Effectiveness Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not at all | 0
  1 = Slightly | 0
  2 = Somewhat | 1
  3 = Mostly | 5
  4 = Very | 5

24. Primary Outcome: Internet Impact and Effectiveness Questionnaire: Participants Response to "Improvement in Difficulties Falling Asleep"
Description: Participants expressed any improvement in difficulty falling asleep as a result of SHUTi with a survey item on a 5-point scale, "SHUTi helped improve my difficulties with falling asleep" with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Impact and Effectiveness Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not at all | 0
  1 = Slightly | 1
  2 = Somewhat | 2
  3 = Mostly | 2
  4 = Very | 6

25. Primary Outcome: Internet Impact and Effectiveness Questionnaire: Participants Response to "Improvement in Waking up in the Middle of the Night"
Description: Participants expressed any improvement in waking up in the middle of the night as a result of SHUTi with a survey item on a 5-point scale, "SHUTi helped improve my difficulties with waking up in the middle of the night" with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Impact and Effectiveness Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not at all | 0
  1 = Slightly | 4
  2 = Somewhat | 0
  3 = Mostly | 1
  4 = Very | 6

26. Primary Outcome: Internet Impact and Effectiveness Questionnaire: Participants Response to "Improvement in Difficulties Waking up Too Early"
Description: Participants expressed any improvement in difficulties waking up too early as a result of SHUTi with a survey item on a 5-point scale, "SHUTi helped improve my difficulties with waking up too early" with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Impact and Effectiveness Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not at all | 2
  1 = Slightly | 0
  2 = Somewhat | 3
  3 = Mostly | 4
  4 = Very | 2

27. Primary Outcome: Internet Impact and Effectiveness Questionnaire: Participants Response to "Improvement in Sleep Quality"
Description: Participants expressed any improvement in sleep quality as a result of SHUTi with a survey item on a 5-point scale, "SHUTi helped improve my sleep quality" with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Impact and Effectiveness Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not at all | 0
  1 = Slightly | 0
  2 = Somewhat | 2
  3 = Mostly | 3
  4 = Very | 6

28. Primary Outcome: Internet Impact and Effectiveness Questionnaire: Participants Response to "Increase in Insomnia Knowledge"
Description: as for outcome 19
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Impact and Effectiveness Questionnaire. One of 11 participants did not respond to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 10
Participants
  0 = Not at all | 1
  1 = Slightly | 0
  2 = Somewhat | 1
  3 = Mostly | 3
  4 = Very | 5

29. Primary Outcome: Internet Impact and Effectiveness Questionnaire: Participants Response to "Improvement in Daytime Functioning"
Description: Participants expressed any improvement in daytime functioning as a result of SHUTi with a survey item on a 5-point scale, "SHUTi helped improve aspects of my daytime functioning like alertness, performance, work attendance, etc." with '0= not at all' to '4=very'
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Impact and Effectiveness Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not at all | 0
  1 = Slightly | 2
  2 = Somewhat | 2
  3 = Mostly | 3
  4 = Very | 4

30. Primary Outcome: Internet Intervention Adherence Questionnaire: Participants Response to "Tablet as a Primary Device Used to Access SHUTi"
Description: Participants responded to using tablet as the primary device to access SHUTi with a survey item, "Did you primarily use the tablet to access SHUTi?" with a "yes or no" response
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Intervention Adherence Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = No | 1
  1 = Yes | 10

31. Primary Outcome: Internet Intervention Adherence Questionnaire: Participants Response to "Working Internet Connection"
Description: Participants responded to internet connection problems with a survey item with four options, "My internet connection did not work" with 0 = Not a problem, 1 = A little problem 2 = A major problem, & N/A (Not applicable)
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Intervention Adherence Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not a problem | 8
  1 = A little problem | 0
  2 = A major problem | 1
  N/A (Not applicable) | 2

32. Primary Outcome: Internet Intervention Adherence Questionnaire: Participants Response to Connection Problem to SHUTi
Description: Participants responded to SHUTi connection problems with a survey item with four options, "My internet connection worked, but I could not get connected to SHUTi" with 0 = Not a problem, 1 = A little problem 2 = A major problem, & N/A (Not applicable)
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Intervention Adherence Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not a problem | 7
  1 = A little problem | 0
  2 = A major problem | 0
  N/A (Not applicable) | 4

33. Primary Outcome: Internet Intervention Adherence Questionnaire: Participants Response to "Slow Internet Connection"
Description: Participants responded to slow internet connection with a survey item with four options, "My internet connection was too slow; SHUTi seemed to 'hang'" with 0 = Not a problem, 1 = A little problem 2 = A major problem, & N/A (Not applicable)
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Intervention Adherence Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not a problem | 5
  1 = A little problem | 1
  2 = A major problem | 0
  N/A (Not applicable) | 5

34. Primary Outcome: Internet Intervention Adherence Questionnaire: Participants Response to "Problems With Device"
Description: Participants responded to device problems with a survey item with four options, "My device wasn't working or was having problems" with 0 = Not a problem, 1 = A little problem 2 = A major problem, & N/A (Not applicable)
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Intervention Adherence Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not a problem | 6
  1 = A little problem | 2
  2 = A major problem | 0
  N/A (Not applicable) | 3

35. Primary Outcome: Internet Intervention Adherence Questionnaire: Participants Response to "Forgetting to Access SHUTi"
Description: Participants responded to forgetting to access SHUTi with a survey item with four options, "I just forgot to go to SHUTi" with 0 = Not a problem, 1 = A little problem 2 = A major problem, & N/A (Not applicable)
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Intervention Adherence Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not a problem | 3
  1 = A little problem | 6
  2 = A major problem | 0
  N/A (Not applicable) | 2

36. Primary Outcome: Internet Intervention Adherence Questionnaire: Participants Response to "Not Wanting to Access SHUTi"
Description: Participants responded to not wanting to access SHUTi with a survey item with four options, "I didn't want to go to SHUTi" with 0 = Not a problem, 1 = A little problem 2 = A major problem, & N/A (Not applicable)
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Intervention Adherence Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not a problem | 5
  1 = A little problem | 1
  2 = A major problem | 1
  N/A (Not applicable) | 4

37. Primary Outcome: Internet Intervention Adherence Questionnaire: Participants Response to "Personal Issues Interfering With SHUTi Use"
Description: Participants responded to personal issues interfering with SHUTi with a survey item with four options, "Personal issues stopped me from using SHUTi" with 0 = Not a problem, 1 = A little problem 2 = A major problem, & N/A (Not applicable)
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Intervention Adherence Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not a problem | 4
  1 = A little problem | 3
  2 = A major problem | 1
  N/A (Not applicable) | 3

38. Primary Outcome: Internet Intervention Adherence Questionnaire: Participants Response to "Work Issues Interfering With SHUTi Use"
Description: Participants responded to work issues interfering with SHUTi with a survey item with four options, "Work issues stopped me from using SHUTi" with 0 = Not a problem, 1 = A little problem 2 = A major problem, & N/A (Not applicable)
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Intervention Adherence Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not a problem | 5
  1 = A little problem | 1
  2 = A major problem | 1
  N/A (Not applicable) | 4

39. Primary Outcome: Internet Intervention Adherence Questionnaire: Participants Response to "Difficulty Navigating SHUTi"
Description: Participants responded to difficulty navigating SHUTi with a survey item with four options, "SHUTi was too hard to navigate" with 0 = Not a problem, 1 = A little problem 2 = A major problem, & N/A (Not applicable)
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Intervention Adherence Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not a problem | 8
  1 = A little problem | 0
  2 = A major problem | 0
  N/A (Not applicable) | 3

40. Primary Outcome: Internet Intervention Adherence Questionnaire: Participants Response to "Difficulty Understanding SHUTi Content"
Description: Participants responded to difficulty understanding SHUTi content with a survey item with four options, "The SHUTi material was too difficult to understand" with 0 = Not a problem, 1 = A little problem 2 = A major problem, & N/A (Not applicable)
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Intervention Adherence Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not a problem | 8
  1 = A little problem | 0
  2 = A major problem | 0
  N/A (Not applicable) | 3

41. Primary Outcome: Internet Intervention Adherence Questionnaire: Participants Response to "SHUTi Not Being Useful"
Description: Participants responded to SHUTi not being useful with a survey item with four options, "The SHUTi program did not seem very useful" with 0 = Not a problem, 1 = A little problem 2 = A major problem, & N/A (Not applicable)
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Intervention Adherence Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not a problem | 8
  1 = A little problem | 0
  2 = A major problem | 0
  N/A (Not applicable) | 3

42. Primary Outcome: Internet Intervention Adherence Questionnaire: Participants Response to SHUTi Program Being Too 'Wordy'
Description: Participants responded to SHUTi program being too wordy with a survey item with four options, "The SHUTi program had too many words" with 0 = Not a problem, 1 = A little problem 2 = A major problem, & N/A (Not applicable)
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Intervention Adherence Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not a problem | 8
  1 = A little problem | 0
  2 = A major problem | 0
  N/A (Not applicable) | 3

43. Primary Outcome: Internet Intervention Adherence Questionnaire: Participants Response to Screen Being Too Hard to Read
Description: Participants responded to screen being hard to read with a survey item with four options, "The screen has hard to read (e.g. words were too small)" with 0 = Not a problem, 1 = A little problem 2 = A major problem, & N/A (Not applicable)
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Intervention Adherence Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not a problem | 8
  1 = A little problem | 0
  2 = A major problem | 0
  N/A (Not applicable) | 3

44. Primary Outcome: Internet Intervention Adherence Questionnaire: Participants Response to "Too Much to do in SHUTi"
Description: Participants responded to having too much to do in SHUTi with a survey item with four options, "The daily requirements were too much for me to do" with 0 = Not a problem, 1 = A little problem 2 = A major problem, & N/A (Not applicable)
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Intervention Adherence Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not a problem | 7
  1 = A little problem | 2
  2 = A major problem | 0
  N/A (Not applicable) | 2

45. Primary Outcome: Internet Intervention Adherence Questionnaire: Participants Response to "Diaries Taking Too Long to Complete"
Description: Participants responded to diaries took too long with a survey item with four options, "The diaries took too long to complete" with 0 = Not a problem, 1 = A little problem 2 = A major problem, & N/A (Not applicable)
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Intervention Adherence Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not a problem | 8
  1 = A little problem | 0
  2 = A major problem | 1
  N/A (Not applicable) | 2

46. Primary Outcome: Internet Intervention Adherence Questionnaire: Participants Response to "SHUTi Helping With Insomnia"
Description: Participants responded to SHUTi helping with insomnia with a survey item with four options, "I didn't think SHUTi was really going to help" with 0 = Not a problem, 1 = A little problem 2 = A major problem, & N/A (Not applicable)
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Intervention Adherence Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not a problem | 3
  1 = A little problem | 5
  2 = A major problem | 1
  N/A (Not applicable) | 2

47. Primary Outcome: Internet Intervention Adherence Questionnaire: Participants Response to "Too Many Sleep Rules"
Description: Participants responded to too many sleep rules with SHUTi with a survey item with four options, "There were too many sleep rules to follow" with 0 = Not a problem, 1 = A little problem 2 = A major problem, & N/A (Not applicable)
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Intervention Adherence Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not a problem | 6
  1 = A little problem | 2
  2 = A major problem | 0
  N/A (Not applicable) | 3

48. Primary Outcome: Internet Intervention Adherence Questionnaire: Participants Response to "Spouse/Significant Other/Roommate Having Issues With Participant Using SHUTi"
Description: Participants responded to spouse/significant other/roommate having issues with participants using SHUTi with a survey item with four options, "My spouse/significant other/roommate did not like me using SHUTi or following the sleep rules" with 0 = Not a problem, 1 = A little problem 2 = A major problem, & N/A (Not applicable)
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Intervention Adherence Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not a problem | 3
  1 = A little problem | 1
  2 = A major problem | 0
  N/A (Not applicable) | 7

49. Primary Outcome: Internet Intervention Adherence Questionnaire: Participants Response to "Difficulty With Sleep Restriction Instructions"
Description: Participants responded to difficulty with sleep restriction with a survey item with four options, "I could not stick to the sleep restriction instructions" with 0 = Not a problem, 1 = A little problem 2 = A major problem, & N/A (Not applicable)
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Intervention Adherence Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not a problem | 4
  1 = A little problem | 4
  2 = A major problem | 1
  N/A (Not applicable) | 2

50. Primary Outcome: Internet Intervention Adherence Questionnaire: Participants Who Responded to "Sleep Efficiency Not Improving"
Description: Participants responded to sleep efficiency not improving with a single categorical survey statement, "My sleep efficiency was not improving" on a 4-point Likert scale
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Intervention Adherence Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not a problem | 6
  1 = A little problem | 1
  2 = A major problem | 0
  -88 = N/A (Not applicable) | 4

51. Primary Outcome: Internet Intervention Adherence Questionnaire: Participants Response to "Too Much Homework"
Description: Participants responded to too much homework with SHUTi with a survey item with four options, "There was too much homework" with 0 = Not a problem, 1 = A little problem 2 = A major problem, & N/A (Not applicable)
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Intervention Adherence Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not a problem | 8
  1 = A little problem | 0
  2 = A major problem | 0
  N/A (Not applicable) | 3

52. Primary Outcome: Internet Intervention Adherence Questionnaire: Participants Response to "Homework Difficulty"
Description: Participants responded to homework being too difficult with a survey item with four options, "The homework was too difficult" with 0 = Not a problem, 1 = A little problem 2 = A major problem, & N/A (Not applicable)
Time Frame: 9-11 Weeks post SHUTi initiation
Population: The analysis included participants who completed the Internet Intervention Adherence Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 11
Participants
  0 = Not a problem | 7
  1 = A little problem | 0
  2 = A major problem | 0
  N/A (Not applicable) | 4

53. Primary Outcome: Average Login Counts
Description: SHUTi system generated report of each participant's login counts while they had access to the web based SHUTi program 6-7 months after discharge from inpatient admission
Time Frame: 6-7 months post discharge from inpatient admission for this study
Population: This include all participants who started SHUTi
Measure: Mean (Standard Deviation); unit: Logins
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 25
Logins | 46.36 (41.51)

54. Primary Outcome: Mean Diary Completion Counts
Description: SHUTi system generated report of each participant's number of completed diaries while they had access to the web based SHUTi program 6-7 months after discharge from inpatient admission
Time Frame: 6-7 months post discharge from inpatient admission for this study
Population: This include all participants who started SHUTi
Measure: Mean (Standard Deviation); unit: Count of Diary Completion
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 25
Count of Diary Completion | 65.6 (30.90)

55. Primary Outcome: Average Number of Sessions Completed
Description: SHUTi system generated report of each participant's number of completed sessions during the 9-11 week period after starting the first SHUTi session
Time Frame: 9-11 Weeks post SHUTi initiation
Population: This include all participants who started SHUTi
Measure: Mean (Standard Deviation); unit: Count of sessions completed
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
Number analyzed (Participants) | 25
Count of sessions completed | 4.35 (2.25)

ADVERSE EVENTS:
Time Frame: 9-11 weeks while actively completing the sessions
Arm/Group | Feasibility and Acceptability of Sleep Healthy Using the Internet (SHUTi) for CBT-I
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/58/NCT03493958/Prot_SAP_000.pdf